CLINICAL TRIAL: NCT06567392
Title: Phase I Clinical Trial of Mass Balance of [14C] HRS-5965 in Healthy Chinese Subjects
Brief Title: A Study to Evaluate the Mass Balance of [14C] HRS-5965 in Healthy Adult Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chengdu Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HRS-5965-105
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Complement Mediated Primary or Secondary Glomerular Diseases

STUDY DESIGN:
Intervention Model Description: Single oral dose of [14C] HRS-5965
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C] HRS-5965 (Experimental)
  Interventions: Drug: [14C] HRS-5965

INTERVENTIONS:
Drug: [14C] HRS-5965 — Patients will receive single dose of orally [14C] HRS-5965 on Day 1.

SUMMARY:
Evaluate the Mass Balance of [14C] HRS-5965 in Healthy Adult Volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form prior to the trial and have a full understanding of the trial's procedures, content, and potential adverse reactions;
2. Healthy adult males between 18 and 45 years;
3. Body weight ≥50 kg, and the body mass index (BMI) of 19 to 26 kg/m2;
4. From the signing of the informed consent form until 12 months after the last administration, the subject (including partner) has no family planning and is willing to use the high-efficiency contraceptive measures specified in the plan.

Exclusion Criteria:

1. Comprehensive physical examination, vital signs, laboratory tests (blood routine, blood biochemistry, coagulation function, urine analysis, fecal analysis, thyroid function), full chest anteroposterior and lateral film, abdominal ultrasound, and anoscope results that the researcher deems clinically significant.
2. Patients with QTcF>450 msec at the time of screening or baseline, or 12 lead electrocardiogram examination are abnormal and determined by the researcher to have clinical significance.
3. Patients with clinically significant abnormalities in ophthalmic examinations (color vision, slit lamp, intraocular pressure, and fundus photography).
4. Patients whose blood creatinine levels exceed the upper limit of normal values.
5. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) exceeding the upper limit of normal values (ULN), or total bilirubin exceeding 1.5 times ULN.
6. Hepatitis B surface antigen (HBsAg) positive, or anti hepatitis C virus (HCV) antibody positive, or human immunodeficiency virus (HIV) antibody positive, or Treponema pallidum antibody positive.
7. Abuse of drugs or use of soft drugs (such as marijuana) in the three months prior to screening, or use of hard drugs (such as amphetamines, phencyclidine, etc.) in the year prior to screening; Or screening period urine drug test positive individuals.
8. Patients used any drugs (including prescription drugs, over-the-counter drugs, Chinese herbal medicines, traditional Chinese patent medicines and simple preparations and dietary supplements) within 4 weeks before screening; Or select those who are within 5 half-lives of the drug at the time of screening (whichever is longer).
9. Patients who are allergic to two or more allergens, or who have been determined by the researcher to be potentially allergic to the investigational drug or its components 11. Any clinical history of serious diseases or conditions that the researcher believes may affect the trial results, including but not limited to a history of circulatory, endocrine, nervous, digestive, urinary, or blood, immune, mental, and metabolic diseases.
10. According to the judgment of researchers, there may be diseases or medical conditions that may affect drug absorption, distribution, metabolism, and excretion, or may reduce compliance.
11. Patients with combined diseases of the respiratory, circulatory, digestive, urinary, psychiatric, hematological, endocrine, metabolic, and immune systems.
12. Patients with a history of meningococcal infection or first-degree relatives with a history of meningococcal infection.
13. Screening for individuals with clear evidence of infection (positive pathogen test or previous systemic antibiotic treatment) or those with a body temperature above 38 ℃ within the first 2 weeks.
14. Screening for individuals with severe trauma or surgery within the first 8 weeks, or those planning to undergo surgery during the trial period.
15. Subjects with a history of recurrent oral ulcers.
16. Perianal diseases with hemorrhoids or periodic/ongoing rectal bleeding; The subject is unable to swallow or has difficulty swallowing, or has a history of gastrointestinal dysfunction such as irritable bowel syndrome, inflammatory bowel disease, or has undergone surgery such as gastrectomy, which the researcher determines may affect drug absorption.
17. Habitual constipation or diarrhea, irregular or difficult bowel movements, or other situations that have been evaluated by the researcher and affect the collection of fecal samples.
18. Have a history of severe vomiting.
19. Screening for individuals who smoke an average of 5 or more cigarettes per day within the first 4 weeks, or who are unable to quit nicotine containing products (including nicotine patches) during the trial period.
20. The average daily intake of alcohol in the four weeks before screening exceeds 15 g (15 g of alcohol is equivalent to 450 mL of beer, 150 mL of wine or 50 mL of low alcohol Baijiu), or the alcohol breath test is positive during screening, or the patient uses or drinks any food or drink containing alcohol within 48 hours before administration, or cannot quit during the test.
21. Habitually drinking grapefruit or grapefruit juice or orange juice, or products containing caffeine or xanthine (such as coffee, tea, cola drinks, and chocolate), or using these products within 48 hours before administration, or unable to quit during the trial period.
22. Clinical trials involving any other drug or medical device within the first 3 months of screening or planned to be conducted during the study period, or those who are still within 5 half-lives of the drug before screening (whichever is longer).
23. Vaccines administered within 2 weeks prior to the first administration or planned during the study period and within 1 month after the last administration.
24. Individuals with a history of blood donation or severe blood loss (blood loss ≥ 400 mL) within the 8 weeks prior to screening, or those who have received a blood transfusion within the 12 weeks prior to screening.
25. Engaged in workers who require long-term exposure to radioactive conditions; Or select individuals who have had significant radiation exposure (chest/abdominal CT ≥ 2 times, or other types of X-ray examinations ≥ 3 times) or participated in radiopharmaceutical labeling trials within the previous year.
26. Difficulty in venous blood collection or inability to withstand blood collection due to physical condition; Or subjects who are expected to be unable to complete the entire trial follow-up.
27. The researcher determined that the subjects had other factors that were not suitable for participation in this study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2024-09-03 (Actual); Primary Completion 2024-10-08 (Actual); Study Completion 2024-10-08 (Actual)

PRIMARY OUTCOMES:
Total radioactive recovery rate in urine and feces at each time interval | 0-240 hours
Cumulative total radioactive recovery rate in urine and feces | 0-240 hours
3. Percentage of parent drug and its metabolites in plasma as a percentage of total radioactive exposure (%AUC) | 0-192 hours
Percentage of parent drug and its metabolites in urine and feces as a percentage of administered dose (%Dose) | 0-240 hours
Radioactivity Tmax | 0-192 hours
Radioactivity Cmax | 0-192 hours
Radioactivity AUC | 0-192 hours
Radioactivity t1/2 | 0-192 hours
Radioactivity CL/F | 0-192 hours
Radioactivity Vz/F | 0-192 hours
Total radioactivity ratio for blood/plasma | 0-96 hours

SECONDARY OUTCOMES:
Plasma HRS-5965: Tmax | 0-192 hours
Plasma HRS-5965: Cmax | 0-192 hours
Plasma HRS-5965: AUC | 0-192 hours
Plasma HRS-5965: t1/2 | 0-192 hours
Plasma HRS-5965: CL/F | 0-192 hours
Plasma HRS-5965: Vz/F | 0-192 hours
Plasma HRS-5965: λz | 0-192 hours
AEs and SAEs | 0-11 days

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital Of Shandong First Medical University（Shandong Provincial Qianfoshan Hospital）, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided